CLINICAL TRIAL: NCT04053985
Title: The Efficacy of Transarterial Chemoinfusion (TAI) Combine Lenvatinib in Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-076-01
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAI+lenvatinib group (Experimental): TAI combine lenvatinib
  Interventions: Combination Product: TAI combine lenvatinib
- lenvatinib group (Active Comparator): lenvatinib only
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Combination Product: TAI combine lenvatinib — TAI combine lenvatinib
  Arms: TAI+lenvatinib group
Drug: Lenvatinib — lenvatinib only
  Arms: lenvatinib group

SUMMARY:
evaluation of the efficacy of transarterial chemoinfusion (TAI) combine lenvatinib in advanced hepatocelllar carcinoma

ELIGIBILITY:
Inclusion Criteria:

older than 18 years old and younger than 75 years; ECOG PS≤1; proven hepatocellular carcinoma according patological examination or EASL/AASLD diagnostic criteria; not previous treated for tumor; unresectable; the lab test could meet: neutrophil count≥2.0×109/L; hemoglobin≥100g/L; platelet count≥75×109/L; serum albumin≥35g/L; total bilirubin<2-times upper limit of normal; ALT<3-times upper limit of normal; AST<3-times upper limit of normal; serum creatine<1.5-times upper limit of normal; PT≤upper limit of normal plus 4 seconds; INR≤2.2; sign up consent

Exclusion Criteria:

cannot tolerate TAI or surgery; known history of other malignancy; be allergic to related drugs; underwent organ transplantation before; be treated before (interferon included); known history of HIV infection; known history of drug or alcohol abuse; have GI hemorrhage or cardiac/brain vascular events within 30 days; pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed up to 60 months
  overall survival
PFS | From date of randomization until the date of progress from any cause, assessed up to 60 months
  progression-free survival

SECONDARY OUTCOMES:
ORR | From date of randomization until the date of death from any cause, assessed up to 60 months
  object response rate
DCR | From date of randomization until the date of death from any cause, assessed up to 60 months
  disease control rate

CONTACTS AND LOCATIONS:
Locations (1):
- SUN YAT-SEN University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided